CLINICAL TRIAL: NCT06329102
Title: Right Colectomy for Colon Cancer Database
Brief Title: Right Colectomy for Colon Cancer Database (RCC). Surgical Technique, Route of Access and Quality of the Specimen
Acronym: RCC
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 93628
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Right Sided Colon Cancer; Right Colectomy; Lymphadenectomy
MeSH Terms: interventions — Minimally Invasive Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Access (Open, laparoscopic, robotic): Outcomes will be analysed for the different groups
  Interventions: Procedure: Surgical access
- Extend of lymphadenectomy described by VAS score: The extend of lymphadenectomy achieved will be described by a visual analogue scale (VAS) after the operation
  Interventions: Procedure: Surgical access
- Quality of the specimen: The quality of the specimen will be documented postoperatively by a graded classification system
  Interventions: Procedure: Surgical access

INTERVENTIONS:
Procedure: Surgical access — Complications by Clavien Dindo Number of lymph nodes. Disease free and Overall survival
  Other Names: Complications, oncological outcome, survival

SUMMARY:
Aim of the project is to surveil results after extended lymphadenectomy for right sided colon resection for cancer with different operative techniques. Patients operated for right sided colon cancer will be involved. There are different operative methods used in terms of extend of lymphadenectomy and access (open, laparoscopic and robotic assisted) that are already implemented. The Norwegian standard operation contains less extended lymph node dissection. Patients operated by the standard method will serve as control group. Choice of access and extend of lymph node dissection in Norway is dependant on the surgeon and hospital. At Haukeland University Hospital extend and access of surgery are determined by a multidisciplinary team meeting. More radical surgery might result in more complications and the benefit for the patients in terms of oncological result and survival is uncertain. At Haukeland University Hospital, extended lymphadenectomy has been mostly performed by open surgery. During the study phase we will introduce extended lymphadenectomy by laparoscopy and robotassisted surgery. Hypothesis is that more radical surgery performed by minimal invasive surgery will result in equal or better oncological results, and less complications, shorter hospital stay and better quality of life. As method we choose a prospective observational study. All eligible patients with adenocarcinoma of the right colon without another ongoing oncological treatment for other cancers will be included. Patientdata will be prospectively registered in a web-based database. Aim of the study will be to define the optimal extend of lymphadenectomy to achieve the best oncological result. In addition, we will analyse the results dependent on the surgical access (open, laparoscopic or robotic). The assumed difference between the operative methods is small. Therefore, the study is designed and approved as a multicenter registration in order to achieve the necessary statistical power.

DETAILED DESCRIPTION:
Right colectomy for colon cancer database

1. Scientific plan: 1.1. Rationale for the project Colon cancer is the third most cancer in Norway. Five-year relative survival for men and women is 65% and 69% respectively. Surgery is the cornerstone of the treatment and about 50% of patients are cured by surgery alone. In 2018, 2117 patients with stage I-III colon cancer were operated in Norway. About half of them with right-sided colectomies. Parallel to the development of minimally invasive surgery, focus on more radical surgical technique has been increasing, inspired by the improved survival in rectal cancer. Despite growing interest in surgical technique, the level of evidence in this area is low. Reasons are the lack of a common definitions of surgical technique and anatomical differences between the right and left colon. There are two sets of terms used to describe radical colon cancer surgery with adequate lymph node harvest and dissection along embryological planes. The Japanese D2 and D3 dissection refers to lymph node stations and the corresponding European "complete mesocolic excision" (CME) and central vascular ligation (CVL) to anatomical planes. Despite the mentioned uncertainties, there is growing evidence that more radical surgery is leading to improved oncological outcome in right- sided colon cancer. Minimal invasive surgery improves quality of life by reducing pain, postoperative complications and thereby reduces hospital stay and convalescence, but there is concern that more radical surgery is associated with more intraoperative injuries and severe non-surgical complications than "conventional" resection for colon cancer. Robotic assisted right-sided colectomy could overcome the technical challenges of more radical surgery with all benefits from minimal invasive surgery. Introduction of new health technologies may cause serious harm to patients and has to be monitored carefully. In Norway, reporting to the Norwegian Cancer Registry and the Norwegian Registry for Gastrointestinal Surgery is mandatory. But both registries do not cover details of the surgical technique, route of access and quality of the specimen.

1.2. Participating institutions and database solution To date, the applicants have several databases approved by the local ethics committee that cover different topics of colorectal cancer. In order to make the database accessible to a larger cohort we decided to create a web-based solution. From the existing databases, a selection of a maximum of 50 parameters have to be transferred.

The database will be designed as an easy to use, cloud-based solution which enables multiuser and multicenter utility. The database will have filters and include tools for analysis and statistics to facilitate generation of descriptive data to be used for data quality assurance and hypotheses testing. This function will also provide regular reports (i.e. every 6 months) to ensure data quality and patient safety during the introduction of more radical surgery and throughout the study. The web-access functionality of the database went through a risk and vulnerability analysis of the local health care authorities and is approved by "Helse Vest IKT". It will also have the possibility to include patient outcome measures (PROMS) and patient reported experience (PREMS) modules. In order to reach statistical power for some hypothesis (i.e. oncological outcome) we will need a sample size that is too big for a single institution. Therefore, the database will be offered to all Norwegian hospitals operating right-sided colectomies.

1.3. Data collection To have a valid control group, all operations for right-sided colon cancer will be registered, including open, laparoscopic and robotic assisted access. The extend of surgery will be documented according to the Japanese D2 and D3 classification, as D2-, complete D2- and D3 dissection. The quality of the specimen will be assessed by the operating surgeon and pathologist by a newly proposed classification system for right-sided colon cancer. Photo documentation of the anatomy after dissection will give the opportunity to analyse the quality of surgery independently. All data will be recorded prospectively immediately after the operation and after 30 days. Long-term outcomes such as survival, hernia, and recurrences shall be checked 6 monthly. In addition, in order to avoid double data entry oncological results will be collected from the Norwegian Cancer Registry and postoperative complications from the Norwegian Registry for Gastrointestinal Surgery. Merging data from national databases is current practice in Norway and there will be no delay. Ethical committee has approved the study. The patients will be asked for informed consent before data collection. Data can be collected in the web-based database Ledidi (Intraoperative, postoperative form) or paper based. Participating other hospitals will get access to the database after signing a collaboration and data processor agreement.

Health related quality of life (HRQoL) is assessed using the 15D instrument (http://www.15d-instrument.net/15d), a validated, standardized, self-administered health state descriptive questionnaire translated into Norwegian that can be used as a profile and single index score measure.

1.4. Database and security: Ledidi Prjcts is a commercially available web-based software solution developed, approved and used by the Oslo University Hospital (Rikshospitalet). The database has been evaluated for risk and security (ROS) and is approved by the local IT provider "Helse Vest IKT".

Ledidi's security system and Prjct's technical architecture are specified and implemented according to requirements and templates from:

* "Normen" (Information security norm in the Norwegian health care sector)
* General Data Protection Regulation (GDPR)
* Health Insurance Portability and Accountability Act
* Strategy, which is the governing perspective

The developers are constantly working to ensure that the technical architecture and security of the solution complies with the requirements referred to above. Ledidi's information security governance consists of:

* Procedures, protection and technology, which constitute the implementing perspective
* Control, to handle nonconformities, among other things Procedures and technical solutions ensure

  1. data integrity and confidentiality, e.g. through a. encryption upon storage and b. encryption during transport
  2. authentication and authorization, implying that only the right people have the right access
  3. 2-factor authentication at login for further verification of user identity
  4. directly identifiable data is only available to users with the correct access level
  5. protection against denial of service attacks (DoS and DDoS) and other types of attacks.
  6. continuous logging and traceability
  7. redundancy and scaling
  8. deletion and return upon requests
  9. secure storage management
  10. backup and restore

1.5. Study Design This is a prospective comparative study, assessing complications and oncological outcome following all types of colectomy procedures for right-sided colon cancer, at the sponsor institution in the first instance. Open, laparoscopic and robotic assisted operations will be included. Data from all patients undergoing the procedures will be collected for at least 3 years in order to obtain information about eventual start of adjuvant chemotherapy, incidence of hernia and oncological outcome (survival, recurrence).

Other institutions will be offered to collect their colectomy data in the Ledidi database for free.

1.6. Aim of the study The primary aim of the project is to compare the impact of surgical radicality on clinical outcomes for right-sided colon cancer. If sufficient sites participate a large sample size could be achieved (see section 2.8), this will also enable statistical comparison of oncological outcomes.

1.7. Study Endpoints Primary endpoint

* Surgical complications (Patient safety) Secondary endpoints
* Surgical quality (Specimen quality, number of lymph nodes)
* Quality of life after surgery
* Oncological outcome (survival, recurrence, adjuvant therapy) Surgical endpoints
* Operating time (min)
* Conversions
* Intraoperative blood loss/ perioperative transfusion units
* Significant incidents of bleeding from superior mesenteric artery, vein or their branches in the mesentery requiring intervention
* Specimen quality
* Reoperations
* Anastomotic leak
* Prolonged postoperative ileus
* Total length of hospital stay/ readmissions within 30 days
* Incisional hernia at 6 months

1.8. Sample Size In Norway, about 1000 right-sided colectomies are performed annually and about 60-80 scheduled, elective procedures at our institution. At present a randomization between to different procedures with different radicality at a single institution will be unethical if the more radical approach is already implemented. For that reason, non-randomization will be the major bias. This could be overcome by multiple centers that stick to detailed definitions of different procedures (D2, D3, complete D3) as mentioned earlier. With a larger sample size, a propensity score in a case control study could be performed. Another possibility will be to compare the results to historical or national data from the registries.

An improvement from 40% complications (Clavian Dindo grade 2-5)14 to 20% in the robotic group is considered statistically significant. To have a 90% power to detect such a difference a sample size of 218 patients is needed. At our hospital about 60- 80 right-sided colectomies were performed annually. Thus, the estimated total accrual period will be 3 years. Regarding oncological results, to show a 10% improvement in 5 years relative survival between standard lymph node dissection (D2) and extended dissection (D3) with a= 0,05 and power of 0,80 will require 555 patients in each arm.

2. Ethical considerations All surgical techniques are used in clinical practice as recommended and defined by national guidelines. But the distribution of access (open or laparoscopic) and the extend of lymph node dissection varies between the different surgeons and the Norwegian hospitals. At Haukeland University Hospital, open D3 dissection has been performed since 2015 and is currently under evaluation by a randomized trial (REK Ref.nr.: 2015/2396: Open D3 right hemicolectomy compared to laparoscopic CME for right sided colon cancer). The study results are published. Robotic assisted right-sided colectomy with extended lymphadenectomy is performed since 2016. Laparoscopic right-sided colectomy is the standard procedure. Since all operative techniques are implemented, the project should not cause ethical problems. But at present, for operations outside a study protocol, the extend of lymph node dissection for right-sided colectomies is not reported. Though a comparison regarding the extend of lymphadenectomy is not possible.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant tumor of the right colon at CT and/or colonoscopy.
* Confirmed adenocarcinoma
* Patients medically cleared by anesthesiologist for general anesthesia and oncological radical resection
* Informed consent

Exclusion Criteria:

* Patients under 18 years
* Patients with recurrent cancer after previous surgery
* Patients with ongoing treatment due to other cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with confirmed adenocarcinom of the right colon admitted to the hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Surgical complications defined by Calvien Dindo II to V | From the operation to discharge and readmission within 30 days
  The primary aim of the project is to compare the impact of surgical radicality on clinical outcomes for right-sided colon cancer. The Clavien Dindo classification is a validated system ranging from I-V.

SECONDARY OUTCOMES:
Surgical quality described by the specimen quality and number of lymph nodes harvested | Postoperatively
  Specimen quality will be assessed by the surgeon postoperatively by a validated classification system for complete mesocolic excision in right-sided colon cancer (Benz S et al) and the number of lymph nodes
Oncological quality will be measured by overall survival and recurrence | Postoperatively up to five years
  Data will be collected from the patient chart up to 5 years after operation
Quality of life after surgery measured with the 15D instrument | 2021 to 2024
  The QoL questionnaire 15D instrument by Sintonen is a validated self-reported instrument. The 15D is a generic, comprehensive, 15-dimensional, standardized, self-administered measure of health-related quality of life (HRQoL) that can be used both as a profile and single index score measure.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Pfeffer, Prof, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Yes
All IPDs that underline results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2024-2024
Access Criteria: signed cooperation agreement
URL: https://app.ledidi.no/login

REFERENCES:
- [Background] Lygre KB, Eide GE, Forsmo HM, Dicko A, Storli KE, Pfeffer F. Complications after open and laparoscopic right-sided colectomy with central lymphadenectomy for colon cancer: randomized controlled trial. BJS Open. 2023 Jul 10;7(4):zrad074. doi: 10.1093/bjsopen/zrad074. PMID 37643373
- [Background] Lygre KB, Eide GE, Liedenbaum MH, Augland IMB, Haldorsen IS, Pfeffer F. Short and equal vascular stump length after standardized laparoscopic and open surgery with central lymphadenectomy for right-sided colon cancer. Br J Surg. 2024 Jan 3;111(1):znad410. doi: 10.1093/bjs/znad410. No abstract available. PMID 38064678
- [Background] Sintonen H. The 15D instrument of health-related quality of life: properties and applications. Ann Med. 2001 Jul;33(5):328-36. doi: 10.3109/07853890109002086. PMID 11491191
- [Background] Benz S, Tannapfel A, Tam Y, Grunenwald A, Vollmer S, Stricker I. Proposal of a new classification system for complete mesocolic excison in right-sided colon cancer. Tech Coloproctol. 2019 Mar;23(3):251-257. doi: 10.1007/s10151-019-01949-4. Epub 2019 Mar 5. PMID 30838463
- [Derived] Pfeffer F, Kalgraff P, Lygre KB, Nedrebo BS, Forsmo HM. Proposal of a new visual analogue scale to describe the extent of lymphadenectomy in right-sided colectomy for cancer-a prospective observational study. Tech Coloproctol. 2025 Sep 2;29(1):166. doi: 10.1007/s10151-025-03182-8. PMID 40892141